CLINICAL TRIAL: NCT04535089
Title: Opioid Sparing Analgesia: Intraoperative Infusion Dexmedetomidine Versus Lidocaine for Intracranial Surgeries in Children
Brief Title: Opioid Sparing Analgesia: Dexmedetomidine Versus Lidocaine for Intracranial Surgeries in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, lecturer of Anaesthesia ,and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6318
Record Dates: First submitted 2020-08-22; First posted 2020-09-01 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomdine (Active Comparator): IV bolus dose of 0.5ug/kg dexmedetomidine diluted in 10ml saline 1% over 15 minutes followed by continuous infusion of 0.5ug/kg/h
  Interventions: Drug: Dexmedetomidine injection
- lidocaine (Active Comparator): IV bolus dose of 1mg/kg lidocaine 1% over 15 minutes followed by continuous infusion of 1.5mg/kg/h
  Interventions: Drug: Lidocaine Iv

INTERVENTIONS:
Drug: Dexmedetomidine injection — receive IV bolus dose of 0.5 ug/kg dexmedetomidine diluted in 10ml saline 1% over 15 minutes followed by continuous infusion of 0.5 ug/kg/h
  Other Names: precedex
  Arms: dexmedetomdine
Drug: Lidocaine Iv — IV bolus dose of 1mg/kg lidocaine 1% over 15 minutes followed by continuous infusion of 1.5mg/kg/h
  Other Names: xylocaine 1%
  Arms: lidocaine

SUMMARY:
Perioperative pain control is necessary in children as inadequate treatment may lead to progression of perception of pain and development of chronic pain in the future.

Anesthetists tend to adopt approach to perioperative control of pain by non-opioid drugs that mediate pain modulation. Its use as opioid sparing analgesia in different surgeries leading to mixed results.

DETAILED DESCRIPTION:
Site of study:

This study will be carried out in neurosurgical operating rooms of Zagazig University Hospitals.

b. Sample size: A pilot study was done to estimate percent of children need intraoperative fentanyl was (10%) for dexmedetomidine group, and ( 40%) for lidocaine group, at 0.05 α error and 0.2 β error . Sample size was calculated using Open Epi software, is 32 children in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-18 years old.
* Sex: both sexes.
* Physical status: American Society Of Anesthesiologist 1& II.
* Body Mass Index >5 th and < the 85th percentile for age.
* Type of operations: elective intracranial surgeries under general anesthesia.
* Duration of operation < 3 hours.
* Written informed consent from the parent of child

Exclusion Criteria:

* Altered mental state
* Unsuitability for extubation.
* Patients on beta blocker, alpha 2 agonist.
* Patients on pain killer or with known history of allergy to study drugs.
* Hepatic, renal, Cardiovascular and respiratory disease.
* The patient has the right to withdraw from the study at any time without any negative consequence on their medical or surgical treatment plan.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative total fentanyl consumption. | from induction till end of surgery up to 3 hours intraoperative.
  Intraoperative fentanyl 0.5ug/ kg when the heart rate and mean arterial blood pressure of patients increased > 20% from basal measurement after exclusion of other causes.

SECONDARY OUTCOMES:
pain intensity | immediately on arrival to PACU, and at 5, 10, 15 minutes till the child will be discharge from PACU postoperative.
  In the Post Anesthesia Care Unite( PACU), the intensity of pain will be assessed using The Wong-Baker Faces Pain Rating Scale (WBFPS) . The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". The child is instructed to choose the face that best describes their intensity of pain currently being experienced immediately on arrival to PACU, and at 5, 10, 15 mintues till the child will be discharge from PACU. The child will be ready for discharge from PACU when attained an Aldrete score ≥9 and free from pain, nausea and vomiting. Protocol for pain management, IV paracetamol 15mg/kg every 6h. maximum daily dose 60mg/kg not exceeding 2grams.
  Child with WBFPS score > 4 will be treated with nalbuphine 0.1mg/kg as rescue analgesic
level of sedation | up to one hour postoperative
  Assessment of level of sedation by 6-point Pediatric Sedation State Scale (PSSS) in the PACU :The six activity states are as follows:
  State 5: Movement impedes procedure and requires forceful immobilization State 4: Movement requires gentle immobilization for positioning State 3: Facial expression of pain or anxiety State 2: Quiet, not moving, no frown, no verbalization of complaint (ideal state) State 1: Deeply asleep with normal vital signs, but requires airway intervention or assistance (e.g., central or obstructive apnea) State 0: Deeply asleep with abnormal physiologic parameters that require acute intervention (e.g., O2 saturation <90%, hypotension, bradycardia).
Time to first call for rescue analgesic (fentanyl) | up to one hour postoperative
  Child with Wong-Baker Faces Pain Rating Scale (WBFPS) score > 4 will be treated with nalbuphine0.1 mg/kg as rescue analgesic as rescue analgesic. The Wong-Baker Faces Pain Rating Scale (WBFPS) . The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". The child is instructed to choose the face that best describes their intensity of pain currently being experienced
Total amount of nalbuphine consumption | up to twelve hours postoperative
  Total amount of nalbuphine consumption in the first 12 hour postoperative
The duration of Post Anesthesia Care Unite stay | up to 2 hour postoperative
  The child will be ready for discharge from PACU to word when attained modified Aldrete score ≥9, fully conscious and no complaint of pain.
side-effects | up to 12 hour postoperative
  side- effects including hypotension MAP < 60, bradycardia HR < 60b/m.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Faculty of medicine, Zagazig, Egypt